CLINICAL TRIAL: NCT01467427
Title: Safety, Efficacy and Pharmacokinetics of NNC-0156-0000-0009 in Previously Treated Children With Haemophilia B
Acronym: paradigm™5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7999-3774; 2011-000826-31 (EudraCT Number); U1111-1119-5013 (Other: WHO); JapicCTI- 121877 (Registry Identifier: JAPIC)
Record Dates: First submitted 2011-10-31; First posted 2011-11-08 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Congenital Bleeding Disorder; Haemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — nonacog beta pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NNC-0156-000-0009 (Experimental)
  Interventions: Drug: nonacog beta pegol

INTERVENTIONS:
Drug: nonacog beta pegol — A single dose of 40 U/kg will be administered intravenously, i.v. (into the vein) once weekly.
  Other Names: NNC-0156-0000-0009

SUMMARY:
This trial is conducted in Asia, Europe and North America. The aim of the trial is to evaluate safety, efficacy and pharmacokinetics (the exposure of the trial drug in the body) of NNC-0156-0000-0009 (nonacog beta pegol, N9-GP) in previously treated children with Haemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with moderately severe or severe congenital haemophilia B with a Factor IX activity level below or equal to 2% according to medical records
* Age below or equal to 12 years (until patient turns 13 years, at time of inclusion)
* Body weight above or equal to 10 kg
* History of at least 50 exposure days (EDs) to other FIX products
* The patient and/or parent(s)/caregiver are capable of assessing a bleeding episode, keeping an electronic diary (eDiary), capable of conducting home treatment and otherwise able to follow trial procedures

Exclusion Criteria:

* Known history of FIX inhibitors
* Current FIX inhibitors above or equal to 0.6 Bethesda Units (BU)
* Congenital or acquired coagulation disorder other than haemophilia B
* Platelet count below 50,000/mcL at screening
* Alanine aminotransferase (ALT) above 3 times the upper limit of normal reference ranges at screening
* Creatinine level above or equal to 1.5 times above the upper normal limit of normal reference ranges at screening
* Human immunodeficiency virus (HIV) positive, defined by medical records, and with a CD4+ lymphocyte count below or equal to 200/mcL
* Immune modulating or chemotherapeutic medication (except single pulse treatment, inhaled and topical steroids)
* Previous arterial thrombotic events (myocardial infarction and intracranial thrombosis, as defined by medical records)

Ages: 0 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2012-05-16 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (26):
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Colorado Hemophilia & Thrombosis Center, Aurora, Colorado
  - Childrens National Medical Ctr, Washington D.C., District of Columbia
  - University of Miami Hospital & Clinics, Miami, Florida
  - Emory University_Atlanta_1, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - University Of Iowa, Iowa City, Iowa
  - University Of Louisville_Louisville_0, Louisville, Kentucky
  - Johns Hopkins University_Baltimore_3, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospitals And Clinics Of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Univ of NE Med Center_Omaha, Omaha, Nebraska
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - Mount Sinai Medical Center, New York, New York
  - Univ Hosp Cleveland Med Ctr, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children Hemostati Ctr, Dayton, Ohio
  - Univ Oklahoma Sci Ctr OK City, Oklahoma City, Oklahoma
  - Children's Hosptl Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt Hemostasis Thrombosis Clinic, Nashville, Tennessee
  - Children's Medical Center_Dallas, Dallas, Texas
  - Texas Children's Hospital_Houston, Houston, Texas
  - Univ TX Hlth Sci Ctr Houston, Houston, Texas
- Brazil (4):
  - Nucleo de Pesquisa Instituto Pele Pequeno Principe, Curitiba, Paraná
  - Universidade Estadual de Campinas, Campinas, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo
  - Hemorio-Fundarj, Rio de Janeiro
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Clinical Hospital Centre Split, Firule, Paediatric Haem. Dpt, Split, Croatia
- France (3):
  - Ap-Hp-Hopital de Bicetre-1, Le Kremlin-Bicêtre
  - Hôpital de la Timone, Marseille
  - Ap-Hp-Hopital Necker-1, Paris
- Germany (2):
  - Coagulation Research Center, Duisburg
  - Medizinische Hochschule Hannover - Pädiatrische Hämato-, Onko- und Hämostasiologie, Hanover
- Istituto di Medicina Int. A. Bianchi Bonomi Univ. Milano, Milan, MI, Italy
- Japan (3):
  - St. Marianna University School of Medicine Hospital_Pediatrics, Kanagawa
  - Shizuoka Children's Hospital, Hematology-Oncology, Shizuoka
  - Ogikubo Hospital_Pediatries & Blood, Tokyo
- National Blood Centre, Kuala Lumpur, Malaysia
- National Taiwan University Children's Hospital, Taipei, Taiwan
- Necmettin Erbakan University Pediatric Hematology, Konya, Turkey (Türkiye)
- United Kingdom (7):
  - Basingstoke & North Hampshire Hospital - Centre for Haemophilia, Haemostasis and Thrombosis, Basingstoke
  - Birmingham Children's Hospital, Birmingham
  - Leicester Royal Infirmary - Haemostasis & Thrombosis Unit, Leicester
  - Leicester Royal Infirmary, Leicester
  - St Thomas' Hospital - Haemostasis and Thrombosis Centre, London
  - St Thomas' Hospital, London
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordiskdisclosure commitment on novonordisk-trials.com

REFERENCES:
- [Background] Safety, efficacy and pharmacokinetics of nonacog beta pegol (N9-GP) in prophylaxis and treatment of bleeding episodes in previously treated pediatric hemophilia B patients. Carcao M, Zak M, Abdul Karim F, Hanabusa H, Kearney S, Lu M-Y, Persson P, Rangarajan S, Santagostino E. Presented 06-Dec-2014 at the American Society of Hematology - 56th Annual Meeting - held in San Francisco, CA, US (poster #1513)
- [Result] Carcao M, Zak M, Abdul Karim F, Hanabusa H, Kearney S, Lu MY, Persson P, Rangarajan S, Santagostino E. Nonacog beta pegol in previously treated children with hemophilia B: results from an international open-label phase 3 trial. J Thromb Haemost. 2016 Aug;14(8):1521-9. doi: 10.1111/jth.13360. Epub 2016 Jun 22. PMID 27174727
- [Result] Carcao M, Kearney S, Lu MY, Taki M, Rubens D, Shen C, Santagostino E. Long-Term Safety and Efficacy of Nonacog Beta Pegol (N9-GP) Administered for at Least 5 Years in Previously Treated Children with Hemophilia B. Thromb Haemost. 2020 May;120(5):737-746. doi: 10.1055/s-0040-1709521. Epub 2020 May 5. PMID 32369845
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 19 sites that screened participants, 17 sites enrolled participants. The trial was therefore conducted at 17 sites in 8 countries, as follows: Canada: 1 site; Germany: 1 site; Italy: 1 site; Japan: 3 sites; Malaysia: 1 site; Taiwan: 1 site; United Kingdom: 3 sites; United States: 6 sites
Pre-assignment Details: The trial was divided into a 52-week main phase where patients received prophylaxis treatment until 50 EDs (Exposure days), followed by an extension phase.
Groups:
- Younger Children (0-6 Years): Participants received nonacog beta pegol 40 U/kg (units/kilogram) intravenous (I.V.) once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
- Older Children (7-12 Years): Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
Period: Overall Study
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Started | 12 | 13
Completed Main Phase | 11 | 13
Entered Extension Phase | 11 | 11
Completed (Trial) | 6 | 4
Not Completed | 6 | 9
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Not continuing in extension phase | 0 | 2
Not completed — Withdrawal during extension phase,- Non-compliance | 0 | 1
Not completed — Withdrawal during extension phase, Withdrawal criteria | 0 | 2
Not completed — Withdrawal during extension phase, Withdrawal of consent | 2 | 1
Not completed — Withdrawal during extension phase, Other | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Younger Children (0-6 Years); Older Children (7-12 Years): Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
- Total: Total of all reporting groups
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years) | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.1 (1.7) | 9.6 (1.6) | 6.5 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 4 | 4 | 8
  Race: Black or African American | 0 | 1 | 1
  Race: White | 8 | 5 | 13
  Race: Other | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Inhibitory Antibodies Against Coagulation Factor IX (FIX) Defined as Titre Above or Equal to 0.6 Bethesda Units (BU)
Description: Inhibitors were analysed with either the Nijmegen modified factor IX Bethesda assay or a heat/cold Nijmegen modified factor IX Bethesda assay. Number of participants who developed inhibitory antibodies against factor IX are reported.
Time Frame: From week 0 to week 52
Population: Safety analysis set (SAS) included all participants exposed to nonacog beta pegol.
Measure: Count of Participants; unit: Participants
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 12 | 13
Participants | 0 | 0

2. Primary Outcome: Incidence of Inhibitory Antibodies Against Coagulation Factor IX (FIX) Defined as Titre Above or Equal to 0.6 Bethesda Units (BU)
Description: as for outcome 1
Time Frame: From week 52 to End of trial (EOT) (approximately week 544)
Population: Safety analysis set (SAS) included all participants exposed to nonacog beta pegol.
Measure: Count of Participants; unit: Participants
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 12 | 13
Participants | 0 | 0

3. Secondary Outcome: Number of Bleeding Episodes During Prophylaxis
Description: The number of bleeding episodes per participant during routine prophylaxis was assessed using the individual annualised bleeding rates (bleeding episodes per participant per year).
Time Frame: From week 0 to EOT (approximately week 544)
Population: Full analysis set (FAS) included all participants with efficacy data after exposure to nonacog beta pegol.
Measure: Median (Inter-Quartile Range); unit: bleeds/participant/year
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 12 | 13
bleeds/participant/year | 0.33 [0.05 to 0.87] | 0.78 [0.35 to 1.73]

4. Secondary Outcome: Haemostatic Effect of N9-GP in Treatment of Bleeding Episodes by 4-point Categorical Scale for Haemostatic Response (Excellent, Good, Moderate and Poor)
Description: Description of the haemostatic effect of nonacog beta pegol when used for treatment of bleeding episodes was measured and listed according to the four point scale for haemostatic response as below:
  1. Excellent - abrupt pain relief and/or clear improvement in objective signs of bleeding within 8 hours after a single infusion.
  2. Good - noticeable pain relief and/or improvement in signs of bleeding within 8 hours after a single injection.
  3. Moderate - probable or slight beneficial effect within the first 8 hours after the first injection but requiring more than one infusion within 8 hours.
  4. Poor - no improvement, or worsening of symptoms within 8 hours after two injections.
  A success rate was calculated based on counting good or excellent as successes and poor and moderate as failures.
Time Frame: From week 0 to EOT (approximately week 544)
Population: FAS included all participants with efficacy data after exposure to nonacog beta pegol. Here, overall number of participants analysed=participants who experienced bleeding episodes. Number analysed = participants analysed for specific category for this outcome measure.
Measure: Number; unit: percentage of bleeding episodes
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 9 | 12
percentage of bleeding episodes
  Success | 90.3 | 89.5
  Failure | 9.7 | 10.5

5. Secondary Outcome: Incremental Recovery at 30 Minutes (IR30min)
Description: The incremental recovery was calculated by dividing the baseline-subtracted factor IX activity Units per milliliter (U/mL) measured in plasma 30 min after dosing by the dose injected at time 0 expressed as units per kilogram (U/kg) body weight.
Time Frame: Week 0 (30 minutes after first exposure)
Population: FAS included all participants with efficacy data after exposure to nonacog beta pegol. Here, overall number of participants analysed = Participants who were evaluated for this parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (U/mL)/(U/kg)
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 11 | 13
(U/mL)/(U/kg) | 0.015 (7.31) | 0.016 (16.18)

6. Secondary Outcome: Trough Level (Single-dose )
Description: The mean pre-dose factor IX levels was measured with the one-stage clotting assay during the trial. Geometric mean of the lowest activity of factor IX recorded at week 0 (immediately before next dose was given).
Time Frame: Week 0 (one week after first exposure)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/mL
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 11 | 12
U/mL | 0.084 (16.28) | 0.109 (18.89)

7. Secondary Outcome: Terminal Half-life (t1/2)
Description: Terminal half life is presented at week 0, 30 minutes until one week after first exposure.
Time Frame: Week 0 (30 minutes until one week after first exposure)
Population: FAS included all participants with efficacy data after exposure to nonacog beta pegol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 12 | 13
hours | 69.576 (15.79) | 76.323 (25.48)

8. Secondary Outcome: Trough Level (Steady State)
Description: The mean pre-dose factor IX levels was measured with the one-stage clotting assay during the trial. The estimated mean of the lowest activity recorded immediately before next dose was given from week 4 to EOT approximately (week 544). Data is reported for specific age groups in which participants were a part of at any time from week 4 to EOT, not at specific time points assessed from week 4 to EOT. The analysis is based on a mixed model on the log-transformed plasma concentrations with participant as a random effect and the mean trough level is presented back-transformed to the natural scale. Considering the time frame, actual age groups (adolescents and adults) are added for this outcome measure.
Time Frame: From week 4 to EOT (approximately week 544)
Population: FAS included all participants with efficacy data after exposure to nonacog beta pegol.
  Age groups are based on actual age, therefore some participants are represented in multiple columns.
Measure: Mean (95% Confidence Interval); unit: U/mL
Groups:
- Older Children (7-12 Years): Given the long duration of the combined main and extension phase, 10 patients entered older children group (7-12 years) at some point during the extension phase. Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
- Adolescents(13-17 Years): Given the long duration of the combined main and extension phase, there were 14 patients who became adolescents (13-17 year age group) at some point during the extension phase. Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
- Adult (18-70 Years): Given the long duration of the combined main and extension phase, there were 6 patients became adults (18-70 year age group) at some point during the extension phase. Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years) | Adolescents(13-17 Years) | Adult (18-70 Years)
Number analyzed (Participants) | 12 | 23 | 14 | 6
U/mL | 0.146 [0.127 to 0.166] | 0.193 [0.171 to 0.218] | 0.220 [0.192 to 0.252] | 0.316 [0.254 to 0.394]

9. Secondary Outcome: Number of Adverse Events
Description: An adverse event (AE) was any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Here, data is presented for all adverse events (serious adverse events and other adverse events) from week 0 to EOT approximately (week 544). Data is reported for specific Age Groups in which participants were a part of at any time from week 0 to EOT, not at specific time points assessed from week 0 to EOT (approximately week 544). Considering the time frame, actual age groups (adolescents and adults) are added for this outcome measure.
Time Frame: Week 0 to EOT (approximately week 544)
Population: SAS included all participants exposed to nonacog beta pegol. Here, overall number of participants analysed = participants who experienced bleeding episodes. Number analysed = participants analysed for specific category for this outcome measure.
  Age groups are based on actual age, therefore some participants are represented in multiple columns.
Measure: Number; unit: Events
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years) | Adolescents(13-17 Years) | Adult (18-70 Years)
Number analyzed (Participants) | 12 | 23 | 14 | 6
Events | 252 | 342 | 81 | 10

10. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: A SAE was an experience that at any dose resulted in any of the following: death, a life-threatening experience a), In-patient hospitalisation or prolongation of existing hospitalisation b) a persistent or significant disability/incapacity c) a congenital anomaly/birth defect, Important medical events d) that did not result in death, were life-threatening a) or required hospitalization. Here, data is presented from week 0 to EOT (approximately week 544). Data is reported for specific Age Groups in which participants were a part of at any time from week 0 to EOT, not at specific time points assessed from week 0 to EOT (approximately week 544). Considering the time frame, actual age groups (adolescents and adults) are added for this outcome measure.
Time Frame: Week 0 to EOT (approximately week 544)
Population: as for outcome 9
Measure: Number; unit: Events
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years) | Adolescents(13-17 Years) | Adult (18-70 Years)
Number analyzed (Participants) | 12 | 23 | 14 | 6
Events | 3 | 5 | 1 | 0

11. Secondary Outcome: Medical Events of Special Interest (MESI)
Description: The following events were defined as MESIs: -Medication errors concerning trial products, -Administration of wrong drug,
  * Wrong route of administration,
  * Administration of a high dose with the intention to cause harm, e.g. suicide attempt,
  * Administration of an accidental overdose: more than 20 % from the intended dose,
  * Inhibitor formation against factor IX (FIX),
  * Thromboembolic events,
  * Anaphylactic reaction.
  * Allergic reaction including, but not limited to, any acute immunoglobulin E (IgE) mediated reaction or delayed type hypersensitivity.
  Here, data is presented from week 0 to EOT (approximately week 544). Data is reported for specific Age Groups in which participants were a part of at any time from week 0 to EOT, not at specific time points assessed from week 0 to EOT (approximately week 544). Considering the time frame, actual age groups (adolescents and adults) are added for this outcome measure.
Time Frame: Week 0 to EOT (approximately week 544)
Population: as for outcome 9
Measure: Number; unit: Events
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years) | Adolescents(13-17 Years) | Adult (18-70 Years)
Number analyzed (Participants) | 12 | 23 | 14 | 6
Events | 1 | 3 | 5 | 1

12. Secondary Outcome: Development of Host Cell Protein (HCP) Antibodies
Description: Participants were examined for the development of antibodies against HCP. Number of participants who developed antibodies against HCP is presented.
Time Frame: From week 0 to EOT (approximately week 544)
Population: SAS included all participants exposed to nonacog beta pegol.
Measure: Count of Participants; unit: Participants
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 12 | 13
Participants
  Yes | 1 | 0
  No | 11 | 13

13. Secondary Outcome: FIX Consumption Described as Frequency of Dose/kg for Prophylaxis Use for the Treatment of Bleeding Episodes
Description: Consumption of nonacog beta pegol for treatment of bleeding episodes International units per kilogram per year (IU/Kg/year) per participant is presented from week 0 to EOT approximately (week 544). Data is reported for specific Age Groups in which participants were a part of at any time from week 0 to EOT, not at specific time points assessed from week 0 to EOT (approximately week 544). Considering the time frame, actual age groups (adolescents and adults) are added for this outcome measure.
Time Frame: From week 0 to EOT (approximately week 544)
Population: The FAS included all participants with efficacy data after exposure to nonacog beta pegol. Here, overall number of participants analysed = participants who experienced bleeding episodes. Number analysed = participants analysed for specific category for this outcome measure.
  Age groups are based on actual age, therefore some participants are represented in multiple columns.
Measure: Mean (Standard Deviation); unit: IU/kg/year
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years) | Adolescents(13-17 Years) | Adult (18-70 Years)
Number analyzed (Participants) | 12 | 23 | 14 | 6
IU/kg/year | 2209.3 (79.3) | 2324.9 (83.5) | 2257.6 (121.1) | 1959.5 (533.4)

14. Secondary Outcome: FIX Consumption Described as Amount Consumed for the Treatment of Bleeding Episodes
Description: Average dose of nonacog beta pegol for treatment of bleed from start to stop of bleed is presented from week 0 to EOT approximately (week 544) in international units per kilogram per bleed (IU/Kg/bleed). Data is reported for specific Age Groups in which participants were a part of at any time from week 0 to EOT, not at specific time points assessed from week 0 to EOT (approximately week 544). Considering the time frame, actual age groups (adolescents and adults) are added for this outcome measure.
Time Frame: From week 0 to EOT (approximately week 544)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: IU/kg/bleed
Units Other Than Participants: Bleeds
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years) | Adolescents(13-17 Years) | Adult (18-70 Years)
Number analyzed (Participants) | 12 | 23 | 14 | 6
Number analyzed (Bleeds) | 35 | 75 | 32 | 7
IU/kg/bleed | 53.6 (32.2) | 50.1 (19.4) | 84.3 (110.2) | 59.9 (32.7)

15. Secondary Outcome: Number of Doses of FIX Consumed for the Treatment of Bleeding Episodes
Description: Number of doses of FIX consumed for the treatment of bleeding episodes is presented from week 0 to EOT approximately (week 544). Here, data of number of doses of FIX for the treatment of bleeding episodes is reported among all the participants in an arm. Data is reported for specific Age Groups in which participants were a part of at any time from week 0 to EOT, not at specific time points assessed from week 0 to EOT (approximately week 544). Considering the time frame, actual age groups (adolescents and adults) are added for this outcome measure.
Time Frame: From week 0 to EOT (approximately week 544)
Population: as for outcome 13
Measure: Number; unit: Doses of FIX
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years) | Adolescents(13-17 Years) | Adult (18-70 Years)
Number analyzed (Participants) | 12 | 23 | 14 | 6
Doses of FIX | 1768 | 4201 | 2740 | 747

16. Secondary Outcome: Area Under the Curve Activity Versus Time Profile From Time Zero to 168 Hours Post Dose (AUC(0-168))
Description: Area under the curve activity versus time profile from time zero to 168 hours post dose of nonacog beta pegol is presented.
Time Frame: 0-168 hours post-dosing at week 0
Population: The FAS included all participants with efficacy data after exposure to nonacog beta pegol.
Measure: Mean (Standard Deviation); unit: Units*hour per milliliter (U*h/mL)
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 12 | 13
Units*hour per milliliter (U*h/mL) | 37.764 (4.586) | 44.192 (7.300)

17. Secondary Outcome: Clearance (CL)
Description: Clearance of nonacog beta pegol after single dose is presented.
Time Frame: 0-168 hours post-dosing at week 0
Population: The FAS included all participants with efficacy data after exposure to nonacog beta pegol.
Measure: Mean (Standard Deviation); unit: Milliliters/hour/kilogram (mL/h/kg)
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 12 | 13
Milliliters/hour/kilogram (mL/h/kg) | 0.764 (0.102) | 0.664 (0.147)

18. Secondary Outcome: Mean Residence Time (MRT)
Description: Mean residence time (MRT) of nonacog beta pegol after single dose is presented.
Time Frame: 0-168 hours post-dosing at week 0
Population: The FAS included all participants with efficacy data after exposure to nonacog beta pegol.
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 12 | 13
Hour (h) | 96.332 (12.995) | 108.16 (29.937)

19. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution at steady state (Vss) of nonacog beta pegol is presented.
Time Frame: 0-168 hours post-dosing at week 0
Population: The FAS included all participants with efficacy data after exposure to nonacog beta pegol.
Measure: Mean (Standard Deviation); unit: Milliliters per kilogram (mL/kg)
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 12 | 13
Milliliters per kilogram (mL/kg) | 73.046 (10.843) | 69.752 (15.253)

20. Secondary Outcome: FIX Activity at 30 Minutes (C30min) (Single Dose)
Description: FIX activity (international units per milliliter (IU/mL)) at 30 minutes after single dose is presented.
Time Frame: 30 min post-dosing at week 0
Population: The FAS included all participants with efficacy data after exposure to nonacog beta pegol. Here, overall number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 11 | 13
IU/mL | 0.544 (0.040) | 0.600 (0.074)

21. Secondary Outcome: FIX Activity at 30 Minutes (C30min) (Steady State)
Description: Mean FIX activity at 30 minutes post-dosing from week 4 to EOT approximately (week 544) (C30min) (steady state) is presented.
Time Frame: 30 min post-dosing from week 4 to EOT (approximately week 544)
Population: The FAS included all participants with efficacy data after exposure to nonacog beta pegol.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 12 | 13
IU/mL | 0.174 [0.146 to 0.208] | 0.197 [0.166 to 0.234]

22. Secondary Outcome: TNO-AZL Preschool Quality of Life (TAPQOL)
Description: The Dutch institute of Prevention and Health and the Leiden University Hospital (TNO-AZL) preschool quality of life clustered into 12 multi-item scales is used to assess the health-related quality of life, such as children's motor, communication, emotions, and body structure. Suitable for children from 6 months to 6 years old (TAPQOL). Parents fill in according to the child's condition. Higher score (range 0-100) represents better outcome. The scale range for each of 12 multi-item scales was (0-100) with high score representing better outcome. In this study, the TAPQOL was assessed for children of age 0-3 years.
Time Frame: Screening (Week -6), week 52, week 176 approximately (visit 17)
Population: The FAS included all participants with efficacy data after exposure to nonacog beta pegol. Here, overall number of participants analysed = participants who experienced bleeding episodes. Number analysed = participants analysed for specific category for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Younger Children (0-3 Years): Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
Arm/Group | Younger Children (0-3 Years)
Number analyzed (Participants) | 7
Score on scale
  Screening (week -6) : Sleeping problems | 80.4 (15.3)
  Week 52: Sleeping problems: number analyzed (Participants) | 6
  Week 52: Sleeping problems | 76.0 (15.5)
  Screening (week -6) : Appetite | 91.7 (11.8)
  Week 52: Appetite: number analyzed (Participants) | 6
  Week 52: Appetite | 90.3 (15.2)
  Screening (week -6) : Lung problems | 100.0 (0.0)
  Week 52: Lung problems: number analyzed (Participants) | 6
  Week 52: Lung problems | 93.2 (13.2)
  Screening (week -6) : Stomach problems | 93.0 (12.1)
  Week 52: Stomach problems: number analyzed (Participants) | 6
  Week 52: Stomach problems | 90.3 (15.2)
  Screening (week -6) : Skin problems | 88.1 (17.9)
  Week 52: Skin problems: number analyzed (Participants) | 6
  Week 52: Skin problems | 90.3 (16.3)
  Screening (week -6) : Motor functioning: number analyzed (Participants) | 6
  Screening (week -6) : Motor functioning | 98.0 (4.9)
  Week 52: Motor functioning: number analyzed (Participants) | 6
  Week 52: Motor functioning | 98.0 (4.9)
  Screening (week -6): Social functioning: number analyzed (Participants) | 6
  Screening (week -6): Social functioning | 97.2 (6.9)
  Week 52: Social functioning: number analyzed (Participants) | 6
  Week 52: Social functioning | 97.2 (6.9)
  Screening (week -6) : Problem behavior | 58.1 (40.8)
  Week 52: Problem behavior: number analyzed (Participants) | 6
  Week 52: Problem behavior | 53.7 (29.6)
  Screening (week -6) : Communication: number analyzed (Participants) | 6
  Screening (week -6) : Communication | 92.8 (14.8)
  Week 52: Communication: number analyzed (Participants) | 6
  Week 52: Communication | 87.5 (14.2)
  Screening (week -6) : Anxiety | 76.1 (16.1)
  Week 52: Anxiety: number analyzed (Participants) | 6
  Week 52: Anxiety | 75.0 (22.9)
  Screening (week -6) : Positive mood | 92.9 (18.9)
  Week 52: Positive mood: number analyzed (Participants) | 6
  Week 52: Positive mood | 100.0 (0.0)
  Screening (week -6) : Liveliness | 97.6 (6.4)
  Week 52: Liveliness: number analyzed (Participants) | 6
  Week 52: Liveliness | 100.0 (0.0)
  Approximately week 176: sleeping problem: number analyzed (Participants) | 6
  Approximately week 176: sleeping problem | 89.7 (15.0)
  Approximately week 176: Appetite: number analyzed (Participants) | 6
  Approximately week 176: Appetite | 94.5 (10.1)
  Approximately week 176: Lung problems: number analyzed (Participants) | 6
  Approximately week 176: Lung problems | 97.2 (6.9)
  Approximately week 176: Stomach problems: number analyzed (Participants) | 6
  Approximately week 176: Stomach problems | 83.2 (10.4)
  Approximately week 176: Skin problems: number analyzed (Participants) | 6
  Approximately week 176: Skin problems | 84.7 (20.0)
  Approximately week 176: Motor functioning: number analyzed (Participants) | 6
  Approximately week 176: Motor functioning | 99.0 (2.4)
  Approximately week 176: Social functioning: number analyzed (Participants) | 6
  Approximately week 176: Social functioning | 86.2 (22.1)
  Approximately week 176: Problem behavior: number analyzed (Participants) | 6
  Approximately week 176: Problem behavior | 58.3 (19.3)
  Approximately week 176: Communication: number analyzed (Participants) | 6
  Approximately week 176: Communication | 95.8 (10.2)
  Approximately week 176: Anxiety: number analyzed (Participants) | 5
  Approximately week 176: Anxiety | 80.2 (18.1)
  Approximately week 176: Positive mood: number analyzed (Participants) | 6
  Approximately week 176: Positive mood | 100.0 (0.0)
  Approximately week 176: Liveliness: number analyzed (Participants) | 6
  Approximately week 176: Liveliness | 94.3 (8.8)

23. Secondary Outcome: Number of Participants With Health Economic Impact of N9-GP Treatment Through Characterisation of General Hospitalisation
Description: Number of participants with health economic impact of N9-GP treatment through characterisation of general hospitalisation is presented. Number of participants hospitalised for 0 & 1 day is presented.
Time Frame: From week 0 to EOT (approximately week 544)
Population: The FAS included all participants with efficacy data after exposure to nonacog beta pegol.
Measure: Count of Participants; unit: Participants
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 4 | 5
Participants
  0 Days | 3 | 5
  1 Day | 1 | 0

24. Secondary Outcome: Health Economic Impact of N9-GP Treatment Through Characterisation of Intensive Care Hospitalisation
Description: Health economic impact of N9-GP treatment is presented through number of intensive care hospitalization days.
Time Frame: From week 0 to EOT (approximately week 544)
Population: The FAS included all participants with efficacy data after exposure to nonacog beta pegol. Here, overall number of participants analyzed = number of participants with available data. Number analysed = participants analysed for specific category for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 4 | 5
Days | 0.0 (0.0) | 0.0 (0.0)

25. Secondary Outcome: Health Economic Impact of N9-GP Treatment Through Characterisation of Bleedings Caused Missing School or Studies
Description: Health economic impact of N9-GP treatment through number of days bleedings caused missing school or studies. Number of participants who missed school or studies for 0,1 and 2 days are presented.
Time Frame: From week 0 to EOT (approximately week 544)
Population: The FAS included all participants with efficacy data after exposure to nonacog beta pegol. Here, overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 11 | 13
Participants
  0 days | 9 | 11
  1 day | 1 | 0
  2 days | 1 | 2

26. Secondary Outcome: Health Economic Impact of N9-GP Treatment Through Characterisation of Number of Days Bleedings Caused Using of Mobility Aids
Description: Health economic impact of N9-GP treatment through number of days the patient used mobility aids (wheelchair and/or crutches) is presented.
Time Frame: From week 0 to EOT (approximately week 544)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 11 | 13
Days | 0.4 (0.7) | 1.0 (3.3)

27. Secondary Outcome: Health Economic Impact of N9-GP Treatment Through Characterisation of Number of Days Bleedings Caused Parents to Miss Work
Description: Health economic impact of N9-GP treatment through number of days bleeding caused parents to miss work is presented from week 0 to EOT approximately (week 544).
Time Frame: From week 0 to EOT (approximately week 544)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Younger Children (0-6 Years) | Older Children (7-12 Years)
Number analyzed (Participants) | 11 | 13
Days | 0.3 (0.6) | 0.5 (0.9)

28. Secondary Outcome: Haemophilia-quality of Life (HAEMO-QOL)
Description: Haemophilia quality of life clustered into 11 multi-item scale which is used to assess haemophilia related quality of life such as children's physical health, feeling, family, friends, sport, treatment, dealing with haemophilia, view of a patient. Here, HAEMO-QOL was assessed for the children of age group 8-12 years. The scale range for each of 11 multi-item scale was 0-100 with high scores indicating low quality of life. Multi-item scores and total score were calculated using the following formula: 1/4(Sum of answered items / number of answered items - 1) x 100. HAEMO-QOL scores range from a 0 to 100 scale where high scores (nearing 100) indicate a low quality of life rating.
Time Frame: Screening (week -6), week 52, EOT (approximately week 544)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Younger Children (8-12 Years): Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
Arm/Group | Younger Children (8-12 Years)
Number analyzed (Participants) | 13
Score on scale
  Screening (week -6) : physical health: number analyzed (Participants) | 12
  Screening (week -6) : physical health | 19.8 (19.1)
  Week 52: physical health: number analyzed (Participants) | 12
  Week 52: physical health | 18.2 (17.0)
  EOT approximately week 544: physical health: number analyzed (Participants) | 2
  EOT approximately week 544: physical health | 7.0 (9.9)
  Screening (week -6) : feeling: number analyzed (Participants) | 12
  Screening (week -6) : feeling | 15.5 (19.3)
  Week 52: feeling: number analyzed (Participants) | 12
  Week 52: feeling | 12.8 (22.9)
  EOT approximately week 544: feeling: number analyzed (Participants) | 2
  EOT approximately week 544: feeling | 12.5 (17.7)
  Screening (week -6) : view: number analyzed (Participants) | 12
  Screening (week -6) : view | 25.8 (18.6)
  Week 52: view: number analyzed (Participants) | 12
  Week 52: view | 20.1 (22.5)
  EOT approximately week 544: view: number analyzed (Participants) | 2
  EOT approximately week 544: view | 23.5 (33.2)
  Screening (week -6) : family: number analyzed (Participants) | 12
  Screening (week -6) : family | 25.0 (16.5)
  Week 52: family: number analyzed (Participants) | 12
  Week 52: family | 16.3 (20.4)
  EOT approximately week 544: family: number analyzed (Participants) | 2
  EOT approximately week 544: family | 17.5 (24.7)
  Screening (week -6): friends: number analyzed (Participants) | 12
  Screening (week -6): friends | 54.3 (23.0)
  Week 52: friends: number analyzed (Participants) | 11
  Week 52: friends | 49.0 (22.3)
  EOT approximately week 544: friends: number analyzed (Participants) | 2
  EOT approximately week 544: friends | 43.5 (53.0)
  Screening (week -6) : perceived support: number analyzed (Participants) | 12
  Screening (week -6) : perceived support | 72.5 (26.1)
  Week 52: perceived support: number analyzed (Participants) | 12
  Week 52: perceived support | 71.5 (32)
  EOT approximately week 544: perceived support: number analyzed (Participants) | 2
  EOT approximately week 544: perceived support | 34.5 (48.8)
  Screening (week -6) : others: number analyzed (Participants) | 12
  Screening (week -6) : others | 14.3 (12.5)
  Week 52: others: number analyzed (Participants) | 11
  Week 52: others | 14.5 (17.3)
  EOT approximately week 544: others: number analyzed (Participants) | 2
  EOT approximately week 544: others | 8.5 (12.0)
  Screening (week -6) : sport: number analyzed (Participants) | 12
  Screening (week -6) : sport | 20.8 (19.4)
  Week 52: sport: number analyzed (Participants) | 12
  Week 52: sport | 22.8 (18.7)
  EOT approximately week 544: sport: number analyzed (Participants) | 2
  EOT approximately week 544: sport | 28.0 (26.9)
  Screening (week -6) : dealing: number analyzed (Participants) | 11
  Screening (week -6) : dealing | 56.5 (27.4)
  Week 52: dealing: number analyzed (Participants) | 11
  Week 52: dealing | 49.6 (22.0)
  EOT approximately week 544: dealing: number analyzed (Participants) | 2
  EOT approximately week 544: dealing | 41.5 (53.0)
  Screening (week -6) : treatment: number analyzed (Participants) | 11
  Screening (week -6) : treatment | 34.7 (16.7)
  Week 52: treatment: number analyzed (Participants) | 11
  Week 52: treatment | 25.1 (19.8)
  EOT approximately week 544: treatment: number analyzed (Participants) | 2
  EOT approximately week 544: treatment | 11.0 (0.0)
  Screening (week -6) : total: number analyzed (Participants) | 11
  Screening (week -6) : total | 31.7 (10.1)
  Week 52: total: number analyzed (Participants) | 11
  Week 52: total | 28.0 (12.5)
  EOT approximately week 544: total: number analyzed (Participants) | 2
  EOT approximately week 544: total | 21.5 (26.2)

29. Secondary Outcome: Hemophilia Treatment Satisfaction (HEMO-SAT)
Description: Haemophilia treatment satisfaction change from baseline (screening week -6) to week 176 (visit 17) is presented. The treatment satisfaction of a bleed with N8-GP was assessed using HEMO-SAT assessment tool which contains a questionnaire with 6 domains (Ease and convenience, efficacy, burden, specialist/nurses, centre/hospital, general satisfaction). The scale range for each 6 domains was (0-100) with lower score indicating higher treatment satisfaction. HEMO-SAT was assessed for the children of age group 4-7 years and 8-12 years. Domain score and total score were calculated using following formula - 1/4 (sum of answered items / Number of answered item - 1) x 100. HEMO-SAT scores range from 0-100, where low scores reflecting greater treatment satisfaction.
Time Frame: Screening (Week -6), week 176 (visit 17)
Population: FAS included all participants with efficacy data after exposure to nonacog beta pegol. Here, overall number of participants analysed = participants who experienced bleeding episodes. Number analysed = participants analysed for specific category for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Younger Children (4-7 Years); Older Children (8-12 Years): Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
Arm/Group | Younger Children (4-7 Years) | Older Children (8-12 Years)
Number analyzed (Participants) | 4 | 11
Score on scale
  Ease and convenience | -6.5 (19.4) | -13.4 (16.2)
  Efficacy | -3.8 (21.3) | -14.5 (23.8)
  Burden | -15.8 (16.0) | -8.5 (13.0)
  Specialist/nurses | -1.8 (2.1) | -0.6 (2.1)
  Centre/hospital | 5.0 (13.5) | -2.3 (6.1)
  General satisfaction | -6.3 (12.5) | -3.5 (8.1)

ADVERSE EVENTS:
Time Frame: Week 0 to EOT (approximately week 544).
Description: The analysis was based on safety analysis set. Treatment emergent AEs were defined as AEs occurring after dosing with trial product.
  Data is reported for specific Age Groups in which participants were a part of at any time from week 0 to EOT, not at specific time points assessed from week 0 to EOT.
Groups:
- Younger Children (0 - 6 Years): Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
- Older Children (7 - 12 Years): Given the long duration of the combined main and extension phase, 10 patients entered older children group (7-12 years) at some point during the extension phase. Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
- Adolescents (13 - 17 Years): Given the long duration of the combined main and extension phase, there were 14 patients who became adolescents (13-17 year age group) at some point during the extension phase. Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
- Adults (18 - 70 Years): Given the long duration of the combined main and extension phase, there were 6 patients became adults (18-70 year age group) at some point during the extension phase. Participants received nonacog beta pegol 40 U/kg I.V. once weekly for 52 weeks in main phase and extension phase till end of trial. Bleeding episodes were treated as soon as they were identified. The dose for treatment of an uncomplicated mild/moderate bleeding episode, e.g. a joint bleed, was a single dose of nonacog beta pegol 40 U/kg I.V. Severe bleeding episodes were treated immediately with 80 U/kg.
Arm/Group | Younger Children (0 - 6 Years) | Older Children (7 - 12 Years) | Adolescents (13 - 17 Years) | Adults (18 - 70 Years)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/23 | 0/14 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/12 | 4/23 | 1/14 | 0/6
Other Adverse Events (participants affected / at risk) | 11/12 | 20/23 | 12/14 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger Children (0 - 6 Years) (N=12) | Older Children (7 - 12 Years) (N=23) | Adolescents (13 - 17 Years) (N=14) | Adults (18 - 70 Years) (N=6)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tourette's disorder (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Younger Children (0 - 6 Years) (N=12) | Older Children (7 - 12 Years) (N=23) | Adolescents (13 - 17 Years) (N=14) | Adults (18 - 70 Years) (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (15) | 3 (4) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (3) | 2 (2) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (2) | 2 (3) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (12) | 7 (16) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (23) | 5 (7) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Ear injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 4 (5) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Growing pains (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (9) | 6 (9) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (12) | 3 (4) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (5) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (5) | 3 (5) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (7) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (16) | 2 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Keratouveitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 5 (9) | 3 (8) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 4 (11) | 2 (3) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myringitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 2 (2) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (14) | 4 (17) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nipple disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (4) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (7) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3) | 6 (13) | 2 (2) | 0 (0)
Penile discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 3 (6) | 3 (6) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 (3) | 1 (7) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Product administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (16) | 6 (13) | 2 (2) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (6) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (11) | 1 (1) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 4 (5) | 3 (7) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Sleep terror (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (4) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (6) | 3 (4) | 1 (4) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (4) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Varicella virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (8) | 4 (7) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT01467427/Prot_SAP_000.pdf